CLINICAL TRIAL: NCT02837718
Title: Minimum Effective Volume Of Local Anesthetic İn USG Guided Axillary Approach Brachial Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, necati alper erdoğmuş, Dr, Ankara City Hospital Bilkent
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AnkaranTRH
Record Dates: First submitted 2016-01-17; First posted 2016-07-20 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2018-12

CONDITIONS: Underdosing of Local Anesthetics

STUDY DESIGN:
Intervention Model Description: A total of 55 ASA I-II patients underwent hand surgery operation by administering USG guided-axillary brachial plexus blockage were included in the study. Ulnar, median and radial nerves were seen and the minimum effective LA volume was investigated starting with total 21 ml of %0.5 bupivacain. After accomplishing the blockage, volume was decreased by 0.5 for each nerves. Block administration time, block onset times, anesthesia times and time to first analgesic requirement were recorded.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupivacaine 0,5% Single arm study (Other): Bupivacaine 0,5% Single arm study
  Interventions: Procedure: bupivakain % 0,5

INTERVENTIONS:
Procedure: bupivakain % 0,5 — Bupivacaine 0,5% The study method was a step-up/step-down sequence model where the dose for following patients was determined by the outcome of the preceding block. The starting dose of bupivacaine was 5 mL per nerve. In the case of block failure, the dose was increased by 0.5 mL per nerve. Conversely, block success resulted in a reduction in dose by 0.5 mL per nerve. Each of the three nerves was treated as a separate entity. Dose adjustments were made to each nerve individually. The volume dose was increased in 0.5 mL at every 5 consecutive cases regardless of the result of the previous block in order to minimize bias occurence. A blinded assistant assessed sensory and motor blockade at 5-min intervals up to 30 min.

SUMMARY:
Background Peripheral nerve blocks with use of USG allowed visualisation of the structures and nerves and made the block administrations safe, quick and comfortable. However there are few publications concerning the minimum local anesthetic volume capable of providing blocks. In this study the investigastors aimed to find Minimum Effective Volume Of Local Anesthetic For Ultrasound-Guided Axillary Brachial Plexus Block in hand, elbow and forehand operations.

Materials & Methods A total of 55 ASA I-II patients underwent hand surgery operation by administering USG guided-axillary brachial plexus blockage were included in the study. Ulnar, median and radial nerves were seen and the minimum effective local anesthetic volume was investigated starting with total 21 ml of %0.5 bupivacain. After accomplishing the blockage, volume was decreased by 0.5 for each nerves. Block administration time, block onset times, anesthesia times and time to first analgesic requirement were recorded.

DETAILED DESCRIPTION:
Matherials and Method This randomized, prospective, double-blinded, single-center study was conducted in accordance with the most recent version of the Helsinki Declaration. Approval for the study was granted by the Ankara Numune Research and Training Hospital Ethics Committee. A total of 55 adult patients classified as American Society of Anesthesiologists (ASA) physical status I-II, who were to undergo elective, forearm, wrist or hand surgery were recruited in this trial. Written informed consent was obtained from each patient. Exclusion criteria were patients with coagulopathy, local anesthetic allergy, local infection, any significant neurological, pysychiatric or congnitive disorder, chronic analgesic use, known neuropathies, infection in the injection site or unwillingness of the patient. After arrival in the operating room, an 20-gauge intravenous catheter was placed in the contralateral forearm. Standard monitoring was used throughout the procedure, including non-invasive arterial blood pressure, heart rate, and pulse oximetry. Patients were divided into groups according to their order of arrival and a five-person group was created. İnitial volume of 7 ml. Per nerve(ulnar, median, radial), totaly 21 ml local anesthetic administered in first group(first five patient). İf the success rate of block is three or more in the group, volume was reduced in the next group of 0.5 ml for each nerve. if the success rate is less than three in the group, study is ended. And minimum effective volume was calculated to be statistically.

Block prosedures All the brachial plexus blocks were performed by the same anesthesiologist. The patient is made comfortable in supine position with the arm abducted and the elbow flexed to 90 degrees. After skin and probe preparation, A linear US probe (HFL 38, 6-13MHz) was placed in the transverse plane at the lateral border of pectoralis major muscle to obtain the best view of the brachial plexus. Image quality is optimised with selection of appropriate depth (within 2 cm), focus range (within 1cm) and gain. The structures of interest are very superficial with the pulsating axillary artery localised within 1 cm . Surrounding the axillary artery, one will find the three out of four terminal branches of the brachial plexus: the median (superficial and lateral to the artery), the ulnar (superficial and medial to the artery) and the radial (posterior and lateral or medial to the artery) nerves. A 5 cm needle (21G, Locoplex, Vygon, Ecouen, France) is inserted parallel to the long axis of the transducer from the lateral side. As the needle is in the same plane as an ultrasound beam, the path of the advancement can be visualised in real time as the needle approaches the target nerves. Ideally, the radial nerve should be targeted first, as it lies posterior to artery, in order to prevent displacing the structures of interest to deeper and obscuring the median and ulnar nerves. The musculocutaneous nerve was blocked separately outside the neurovascular bundle with 3 ml %0.5 bupivacaine at all of the patient. We were also worried about the nerve puncture or intraneural injection. In addition, we also confirmed that the location of the needle tip was not in hypoechoic area before each injection. For further safety, we injected 0.5 ml of local anesthetic as a test dose. If the patients complained of paresthesia or pain, or the injection pressure was high, or the spread of local anesthetic was not visualized, investigastors stopped injection, and withdrew the needles and tried again. The investigastors regarded the paresthesia or pain, or high injection pressure as intraneural injection.

The investigator who testing the block is don't know the dose. Sensory block was evaluated for each nerve distribution using ice to test cold sensation, comparing the anaesthetized arm with the contralateral arm, and graded on a three-point scale (0, no difference between sides; 1, some difference between arms but cold still sensed in the blocked arm; 2, no cold sensation in the blocked arm). Motor block for each nerve was evaluated by asking the patient to extend the flexed arm and wrist (radial nerve), flex the wrist and oppose the second and third fingers and thumb (median nerve), flex and oppose fifth finger towards the thumb (ulnar nerve) and was graded as 0, no change; 1, reduced contraction; 2, no contraction. Data were collected every 5 min for the first 60 min, and then 1,2,4,6,8,10,12,18,24 hours. motor and sensory scale, the total value should be higher than 10, if not surgical anesthesia was considered unsuccessful. sensitive block score must be at least five. VAS determination was performed with a scale of numbers between 0 and 10 cm. 1mg/kg tramadol and 15 mg/kg paracetamol IV infusion were administered to patients with a reequirement for additional analgesia (VAS ≥ 4) . The total number of patients who required additional analgesic drugs was noted. During the initial procedures, the operation and postoperatively, patient satisfaction was evaluated as poor (1), moderate (2), good (3) or very good (4).

Statical Analysis Statistical analysis was applied using SPSS 19.0 statistical software.our sample size calculation method is dixon and massey up and down method. According to this account, n = 2 (SD / SEM) ²; n: sample size, SD (standard deviation): The standard deviation, SEM (standard error of mean) is calculated as the standard error of the mean (SD = 5 mL, SEM = 1.0 mL) n were found in 50 patients. For the aplicational errors we add 5 patient (%10 ). A total of 55 patients were included in the study.

The sample size calculation, made by G * Power 3.0.10 statistical software package (effect size (effect size) = 0.4, α = 0.05, degrees of freedom (df) = 48 and 0.85 power (power (1- β)), the number of 50 patients were found to be adequate. However for practical magnification error with a sample of 10% of 55 patients were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* were age over 18 and under 65 years
* informed consent (IC) signed by the patient
* indication for brachial plexus block (anesthesia and analgesia) in candidates forelective hand surgery
* ASA physical status I or II according to the American Society of Anesthesiologists
* body mass index (BMI) <35 kg/m2.

Exclusion Criteria:

* Cognitive impairment or active psychiatriccondition
* İnfection at the blockade puncture site
* Bleeding disorders
* History of local anesthetic allergy
* Pregnancy
* The patients does not want this method .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Minimum effective volume of bupivacain %0.5 | 1 hour
  Ulnar, median and radial nerves were seen and the minimum effective local anesthetic volume was investigated starting with total 21 ml of %0.5 bupivacain. After accomplishing the blockage, volume was decreased by 0.5 for each nerves

SECONDARY OUTCOMES:
first analgesic requirement | 1 day (0,1, 2, 4, 6, 8, 10, 12, 18, 24 hours)
  Time of Visual analogue scale (VAS) over than 4. Measurument starts after operation finish.

IPD SHARING:
Plan to Share IPD: Undecided